CLINICAL TRIAL: NCT02783651
Title: An Observational Study of Patients With Philadelphia Chromosome-negative Relapsed or Refractory Acute Lymphoblastic Leukemia in the US
Brief Title: An Study of Patients With Ph- Chromosome-negative Relapsed or Refractory Acute Lymphoblastic Leukemia in the US
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20150253
Record Dates: First submitted 2016-05-11; First posted 2016-05-26 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Relapsed/Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No treatment 1: It is planned to have 20-30 sites participating on the trial for chart review of approximately 200-235 patients initiating treatment for Philadelphia chromosome-negative (Ph-) Relapsed or Refractory (R/R) Acute Lymphoblastic Leukemia (ALL) between January 2013 and March 2019.
  Interventions: Other: Other
- No Treatment 2: Initial record abstraction will occur at study site with subsequent reviews occurring at the site every 3 months thereafter until study conclusion on March 2020.
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — No intervention other than routine medical care

SUMMARY:
A retrospective chart review study of Philadelphia chromosome-negative R/R ALL patients in the US.

ELIGIBILITY:
Inclusion Criteria

-Medical records of patients initiating treatment for Ph- R/R ALL at participating clinical centers in the US between January 2013 and March 2019 will be eligible for inclusion.

Exclusion Criteria

* Medical records of patients with Ph+ ALL will be excluded.
* If informed consent is required, medical records of patients who do not provide informed consent will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients initiating treatment for Philadelphia chromosome-negative (Ph-) R/R ALL between January 2013 and March 2019 at participating clinical sites in the US
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Treatment patterns in patients with Ph- R/R ALL | 86 months
Drug utilization in patients with Ph- R/R ALL | 86 months
Healthcare resource utilization in patients with Ph- R/R ALL | 86 months

SECONDARY OUTCOMES:
Receipt of allogeneic stem cell transplantation following salvage treatment | 86 Months
Incidence of selected adverse events including cytokine release syndrome, neurologic events, any events resulting in hospitalizations, and other serious adverse events. | 86 Months
Best response to salvage treatment (chemotherapy or blinatumomab) within 8 weeks and within 12 weeks of initiation of salvage treatment. | 12 Weeks
MRD status within 12 weeks of initiation of salvage treatment | 12 Weeks
Overall survival from the time of initiation of salvage treatment | 86 Months
RFS from time remission achieved with salvage treatment | 86 Months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (17):
  - Research Site, Tucson, Arizona
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Chicago, Illinois
  - Research Site, Ames, Iowa
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Hackensack, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com